CLINICAL TRIAL: NCT00262366
Title: Titration Efficacy of Automatic CPAP Versus Fixed CPAP, Following a Prediction Formula in Patients With OSAS
Brief Title: Comparison of Automatic CPAP to Fixed CPAP for OSAS Following a Prediction Formula
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2005/099
Record Dates: First submitted 2005-12-04; First posted 2005-12-06 (Estimated); Last update posted 2007-12-28 (Estimated); Status verified 2007-12

CONDITIONS: Obstructive Sleep Apnea Syndrome
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Comparison of automatic CPAP versus fixed CPAP

SUMMARY:
Comparison of automatic CPAP with fixed CPAP in patients with OSAS

DETAILED DESCRIPTION:
The polysomnography is divided into two parts, randomly assigned:

* in one part, the patient uses the automatic CPAP device in titration mode
* in the other part, the patient uses the CPAP device, in fixed mode according to the prediction formula

ELIGIBILITY:
Inclusion Criteria:

* Patients with proven Obstructive Sleep Apnea Syndrome
* Apnea-hypopnea-index > 20/h
* Awaking index > 30/h

Exclusion Criteria:

* Severe nasal obstruction
* Hypoventilation
* Excessive sleep fragmentation caused by non-respiratory factors
* COPD (FEV1/FVC < 65%)
* CPAP compliance < 3h per night
* Insufficient sleep time (< 2h TST) during one of both parts of the split night CPAP-titration
* Patients needing > 16 mbar CPAP pressures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45
Dates: Start 2005-05; Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Respiratory control expressed by residual number of obstructive and central apneas, hypopneas and snoring
Arousal index
Pressure profile Auto-CPAP (P50, P95 en Pmax)
All outcomes are measured during polysomnography

SECONDARY OUTCOMES:
Pressure adaptation during polysomnography according to body position and sleep stage, pressure variability
Measurements of comfort, subjective evaluation by the patient by questionnaires immediately after polysomnography

CONTACTS AND LOCATIONS:
Overall Officials: Dirk Pevernagie, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital Ghent, Ghent, Belgium

REFERENCES:
- See also: Website of the University Hospital Ghent — http://www.uzgent.be